CLINICAL TRIAL: NCT03502382
Title: Prediction of Leg Length Discrepancy After Unilateral Total Knee Replacement in Varus Deformity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Abanoub Nagaty Wahba, dr., Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: assiut university medical
Record Dates: First submitted 2018-04-11; First posted 2018-04-18 (Actual); Last update posted 2018-04-19 (Actual); Status verified 2018-04

CONDITIONS: Total Knee Replacement
MeSH Terms: interventions — X-Rays

STUDY DESIGN:
Intervention Model Description: Cases of osteoarthritis of the knee with varus deformity undergoing unilateral TKA.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- radilogical (Other): Radiological: standing antero-posterior full-length digital images of the lower extremities
  Interventions: Diagnostic Test: x-ray

INTERVENTIONS:
Diagnostic Test: x-ray — Radiological: standing antero-posterior full-length digital images of the lower extremities

SUMMARY:
To What degree total knee replacement (TKA) affects leg length discrepancy in patients with varus deformity? Varus deformity, the most commonly encountered deformity in patients undergoing TKA is associated with limb alignment and varying degrees of contractures of medial soft tissue structures, laxity of the lateral soft tissue structures, flexion deformity and medial bone erosion at the knee joint .The challenges in performing TKA in a varus arthritic knee include restoration of limb alignment, balancing the medial and lateral soft tissue tension, equalizing flexion and extension gaps and restoring medial bone loss

DETAILED DESCRIPTION:
Limb length discrepancy (LLD)less than 2cm is usually not noticeable and does not require treatment. LLD over 2cm is usually noticed by the individual affected leading to self compensation by walking on the ball of the foot (toe down) or by tilting the pelvis and curving the spine.Untreated LLD can lead to lower back pain and long leg arthritis of the hip LLD and its effects on patient function have been discussed in depth in the literature with respect to hip arthroplasty but there are few studies that have examined the effect on function of limb length discrepancy following TKA.

Improved surgical techniques and rehabilitation protocols have resulted in excellent knee function and range of motion following TKA.

The investigators are aiming from the study to improve functional outcome in patients with knee osteoarthritis undergoing TKA.

ELIGIBILITY:
Inclusion Criteria:

- 1-Cases of osteoarthritis of the knee with varus deformity undergoing unilateral TKA.

2-Cases with previous unilateral TKA undergoing TKA of the other side.

Exclusion Criteria:

* 1-Cases of osteoarthritis of the knee with valgus deformity. 2-Revision total knee replacement cases. 3-Patients with total hip replacement. 4-Extra-articular lower limb deformities. 5-Cases of bilateral TKA done at same setting. 6-Patients with previous knee surgery. 7-Patients with complicated inrta-operative TKA .

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2019-04-30 (Estimated); Study Completion 2019-04-30 (Estimated)

PRIMARY OUTCOMES:
Measuring ofleg length discrepancy before and after unilateral totalknee replacement. | 1 day
  Measuring ofleg length discrepancy before and after unilateral totalknee replacement.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Abdel-Aal, prof., Study Chair — prof. of orthopaedics
Locations (1):
- Assiut University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
the results

REFERENCES:
- [Derived] Khalifa AA, Mullaji AB, Gendy AN, Ahmed AM, Bakr HM, Khalifa YE, Abdelaal AM. Prediction of leg length change (LLC) after correcting varus and flexion deformity in patients undergoing TKA. Eur J Orthop Surg Traumatol. 2021 Aug;31(6):1199-1205. doi: 10.1007/s00590-020-02853-6. Epub 2021 Jan 9. PMID 33423113
- See also: 1. MihalkoWM, Saleh KJ, Krackow KA, Whiteside LA. Soft-tissue balancing during total knee arthroplasty in the varus knee. J Am Acad Orthop Surg. 2009;17:766-74. — https://pdfs.semanticscholar.org/26de/363e5af4230cb80e7146ea7cfb0baad14b85.pdf